CLINICAL TRIAL: NCT00373854
Title: Hypoglycemia and Endothelial Function
Brief Title: Study of How Low Blood Sugar Affects the Way Blood Vessels Work
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Robert Hoffman, Professor, Ohio State University
Other Study IDs: Endo 208
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Hypoglycemia
Keywords: Hypoglycemia; Endothelial function
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: Low blood sugar (hypoglycemia) decreases function of the lining of the blood vessels in normal humans.

This study is designed to explore how hypoglycemia affects the function of the blood vessel lining. This will be determined by measuring blood flow to the arm before and after occlusion of flow. Blood vessel function will be measured before induction of hypoglycemia, during insulin induced hypoglycemia, and after recovery from hypoglycemia. A second study will be done but without hypoglycemia.

DETAILED DESCRIPTION:
Purpose: The purpose of the research is to learn more about how low blood sugar (low blood glucose or hypoglycemia) affects the way the blood vessels work in healthy people. Subjects who participate in this research project must be in good health and taking no medications.

Methods: A screening visit to the Clinical Research Center of the Ohio State University will be used to assess eligibility to participate. The main study consists of two visits to the Clinical Research Center that occur two to four weeks apart. Each of these visits will involve a procedure known as an insulin clamp. This involves giving insulin and sugar water into a vein. The amount of sugar given varies to keep the blood sugar at a predetermined level. For one of the two visits the blood sugar will be low and the other it will be normal. The function of the blood vessels will be measured three times during each study by measuring blood flow before and after stopping blood flow to the arm for 5 min.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* BMI <27 kg/m2

Exclusion Criteria:

* Pregnancy
* Systolic blood pressure >140 mmHg
* Diastolic Blood pressure >90 mg/dl
* Spot daytime urine microalbumin concentration > 20 μg/mg creatinine
* Past or present history of chronic disease (e.g. cancer, hypertension, cardiovascular disease, chronic inflammatory disease) other than diabetes in type 1 diabetic subjects.
* Use of non prescription medications in the past 3 days
* Use of prescription medications in the past 2 weeks

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2005-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Hoffman, MD, Study Chair — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Observational study